CLINICAL TRIAL: NCT00970372
Title: Compulsory Treatment of Alcohol and Drug Dependent Patients and Dual Diagnosis in 5 Counties of Health Region South-East, Norway
Brief Title: Dual-Diagnosis and Compulsory Treatment
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: SSHF_815360
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Substance-Related Disorders; Dual Diagnosis
Keywords: Coercion
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Involuntary patients: Compulsory treated patients according to the Norwegian Social and Welfare Act of 1992. Most patients have dualdiagnosis.
- Voluntary patients: Voluntary patients on the same wards. Most patients have dual-diagnosis.

SUMMARY:
The Norwegian Social and Welfare Act of 1992, opened for compulsory commitment of patients with serious alcohol and drug problems to inpatient care. Clinical research of compulsory committed dual diagnosed patients is to date unavailable and is demanded by the health authorities of Norway. Because there has been limited examination/screening and no post-treatment research efforts on this group of patients, the investigators have limited knowledge of the treatment as well as the patient group. Do compulsory treated patients differ from those voluntarily admitted? Does this type of treatment influence the patients' motivation to change their behaviour, and does the treatment effort lead to positive outcome effects in the long run?

The primary aim is to acquire new and in depth descriptive knowledge about the compulsory treated group of patients according to: Drug dependence, psychiatric and somatic co-morbidity and socio-demographic characteristics, and investigate whether the treatment yields the intended outcomes in terms of improved substance abuse measures.

A second aim is to compare the group with a corresponding group of voluntarily admitted patients within the same wards. A follow-up interview focusing on motivational issues within 6 months post treatment to evaluate the long-term results of the treatment is planned.

A quasi-experimental, prospective case-control study will be conducted. Compulsory committed patients in five counties during a two year period, will be compared to a group of voluntarily admitted patients. The groups will be compared regarding 1) description and screening 2) motivation to change and 3) outcome results after 6 months.

Both official authorities as well as clinical practitioners would benefit from valid Norwegian results and knowledge within this field to form further policies and evidence based best practice for this vulnerable group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with alcohol and substance use disorders
* Estimated premorbid IQ of 70 or higher

Exclusion Criteria:

* Active drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In five counties there are a total of eight beds reserved for compulsory treatment according to the LOST § 6.2 regulation. Of these, four are situated at the Addiction Unit at Sørlandet Hospital (Kristiansand) and four at the Vestfold Clinic, part of the psychiatric section in the county of Vestfold, Tønsberg. It will be necessary to include both sites for two years of inclusion in this study to obtain sufficient samples, as there are only approximately 35 patients in the compulsory committed category annually in this region. All eligible patients compulsory committed to the two wards in Kristiansand and Tønsberg during a twenty-four month period will be asked to participate during their initial assessment.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2008-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Substance use outcomes measured by Europ-ASI Quality of Life | 6 months after discharge

SECONDARY OUTCOMES:
Psychological distress (SCL-90-R) | 6 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Øistein Kristensen, Study Director — Sørlandet Sykehus HF
Locations (1):
- Sorlandet Hospital, Kristiansand, Vest Agder, Norway

REFERENCES:
- [Derived] Opsal A, Kristensen O, Clausen T. Readiness to change among involuntarily and voluntarily admitted patients with substance use disorders. Subst Abuse Treat Prev Policy. 2019 Nov 6;14(1):47. doi: 10.1186/s13011-019-0237-y. PMID 31694664
- [Derived] Pasareanu AR, Vederhus JK, Opsal A, Kristensen O, Clausen T. Mental distress following inpatient substance use treatment, modified by substance use; comparing voluntary and compulsory admissions. BMC Health Serv Res. 2017 Jan 3;17(1):5. doi: 10.1186/s12913-016-1936-y. PMID 28049461